CLINICAL TRIAL: NCT04404322
Title: Ultra - Brief Crisis IPT-A Based Intervention for Suicidal Children and Adolescents (IPT-A-SCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 17-0634 RMC
Record Dates: First submitted 2020-05-04; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-01

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients are referred to SCMC depression and suicide clinic through the ER, outpatient providers or are self-referred. They undergo an initial evaluation and risk assessment. Following initial evaluation, each subject is assigned to one of three study groups, based on clinical considerations. In this stratified randomization system, the most serious acute cases are generally referred to our ultra-short crisis intervention (IPT- A SCI) and the rest are randomized to either one of the three groups: IPT- A SCI, Treatment as usual (TAU) and waiting list (WL). All participants and their parents complete the questionnaires via a secure electronic interface, with the aid of a trained research assistant. Treatment drop-out rates, thus far, seem low and stand at about 11% for the IPT-A SCI and at about 16% for patients who receive TAU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPT A SCI (Experimental): The IPT-A SCI follows the intervention protocol, which includes an intensive phase of 5 weekly 50-minute sessions and 3 follow up personal emails.
  Interventions: Other: IPT A Suicide Crisis Intervention
- Treatment as usual (Active Comparator): TAU patients receive an integrative combination of psychodynamic, supportive and cognitive behavioural therapy, usually lasting between 10-30 weeks.
  Interventions: Other: Treatment As Usual
- wait list (No Intervention): WL patients are monitored by a trained clinician during their waiting period and complete the study questionnaire battery at the parallel time intervals.

INTERVENTIONS:
Other: IPT A Suicide Crisis Intervention — The intervention is comprised of five weekly sessions followed by monthly emails to the patients and their parents over a period of three months. The first session is aimed at introducing the intervention, assessing depression and suicidal risk and building a safety plan. The safety plan consists of a prioritized list of coping strategies that the patient can use when suicidal risk is increased. The second session is focused on reviewing the patient's interpersonal relationships (using the closeness circle and interpersonal inventory) and conceptualizing the interpersonal problem area. Sessions 3-4 focus on developing and practicing interpersonal, emotional and behavioral coping strategies relevant for suicidal risk. Lastly, in session 5, patient and therapist go over the process and main issues which were worked on, emphasizing relapse prevention by going back to the safety plan. First and fifth sessions always involve the parents.
  Arms: IPT A SCI
Other: Treatment As Usual — patients receive an integrative combination of psychodynamic, supportive and cognitive behavioral therapy, usually lasting between 10-30 weeks
  Arms: Treatment as usual

SUMMARY:
To address the critical need in crisis intervention for children and adolescents at suicidal risk the investigators developed an ultra-brief acute crisis intervention, based on Interpersonal Psychotherapy (IPT). The current adaptation of IPT-A is comprised of five weekly sessions, followed by monthly follow-up caring email contacts to the patients and their parents, over a period of three months.

DETAILED DESCRIPTION:
In recent years, suicidal behaviors have shown substantial increase worldwide. This trend is also prominent in Israel and has led to a dramatic increase in mental health treatment demand resulting in long wait times and low treatment acceptance rate. To address the critical need in crisis intervention for children and adolescents at suicidal risk, the investigators developed an ultra-brief acute crisis intervention, based on Interpersonal Psychotherapy (IPT). IPT is an evidence-based intervention for various psychopathologies among different age groups. The current adaptation of IPT-A is comprised of five weekly sessions, followed by monthly follow-up caring email contacts to the patients and their parents, over a period of three months.

ELIGIBILITY:
Inclusion Criteria:

* depression symptoms
* suicidal behavior

Exclusion Criteria:

* acute medical condition
* intellectual disability
* cognitive impairment
* linguistic limitation

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-04-17 (Estimated); Study Completion 2024-04-17 (Estimated)

PRIMARY OUTCOMES:
Suicide Ideation | Change from Baseline to 5 weeks assessment and 4 months assessment
  suicidal ideation [Suicide Ideation Questionnaire (SIQ) (Reynolds, 1987)]
change in Depression | Change from Baseline to 5 weeks assessment and 4 months assessment
  Mood and Feeling Questionnaire (MFQ) (Angold et al., 1995)

CONTACTS AND LOCATIONS:
Overall Officials: Alan APTER, Prof, Principal Investigator — Rabin MC
Locations (1):
- Schneider Children's Medical Center of Israel, Departemnt of Psychological Medicine, Petah Tikva, Israel